CLINICAL TRIAL: NCT01897311
Title: Hypoalgesic Effect of TENS Modulation in Post-Cesarean Pain: A Clinical Trial Controlled and Randomized.
Brief Title: Effect of Modulation of TENS in Pain After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Piauí (Other)
Responsible Party: Principal Investigator, Janaina Mayer de Oliveira Nunes, Assistent teacher, Universidade Federal do Piauí
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0295.0.045.000-11
Record Dates: First submitted 2013-05-24; First posted 2013-07-11 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2013-07

CONDITIONS: Pain
Keywords: cesarean section; pain; transcutaneous electrical nerve stimulation; postpartum period
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- grupo TENS com frequência de 100 Hz (Experimental): TENS application of high frequency (100 Hz, 100 μs)
  Interventions: Device: transcutaneous electrical nerve stimulation
- grupo TENS com frequência de 4 Hz (Experimental): Application of low-frequency TENS (4 Hz, 100 μs)
  Interventions: Device: transcutaneous electrical nerve stimulation
- Placebo with TENS off (Placebo Comparator): TENS application when off
  Interventions: Device: transcutaneous electrical nerve stimulation

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation

SUMMARY:
The aim of the study was to evaluate the analgesic effect of transcutaneous electrical nerve stimulation High (100 Hz) and low (4 Hz) frequency in postpartum pain after cesarean section.

DETAILED DESCRIPTION:
Mothers were randomly divided into three groups (G100, G4 and placebo (GP) - appliance off) and evaluated by NRS (numeric rating scale) before, immediately after application of TENS, and every 20 minutes until he was one hour after the application of electroanalgesia, to verify its effectiveness over time.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years
* present pain at the site of surgical incision less than three according to Category Numerical Scale (NRS)
* literate oriented as to time and space
* with spinal anesthesia before surgery
* incision pfannenstiel type with absence of genitourinary pathology
* primiparous or multiparous

Exclusion Criteria:

* patients with abnormal sensitivity to clinical examination
* demyelinating diseases
* spinal cord injury
* hemorrhage
* infection
* fever
* anesthetic complications
* hypertension, mammary, intolerance, irritation or strong discomfort at the injection site caused by TENS

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Intensity of pain after cesarean | after TENS application

CONTACTS AND LOCATIONS:
Overall Officials: Janaina Mayer de Oliveira Nunes, Principal Investigator — University Federal Piauí
Locations (1):
- Santa Casa de Misericordia Hospital and State Hospital Dirceu Arco Verde, Parnaíba, Piauí, Brazil

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021